CLINICAL TRIAL: NCT02197871
Title: Effects of Nutritional Supplementation in Malnourished Patients in Stable COPD:a Randomised Controlled Trial
Brief Title: Effects of Nutritional Supplementation in Malnourished Patients in Stable COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhujiang Hospital (Other)
Collaborators: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CX20140718
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2014-07-23 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Obstructive Pulmonary Disease(COPD); Malnutrition
Keywords: COPD; malnutrition; nutrition supplementation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- blank control (No Intervention): usual diet
- nutrition supplementation (Experimental): In addition to usual diet,the patients will be given enteral nutrition emulsion, which is a oral nutrition liquid composed of proteins,omega-3 fatty acids,carbohydrate,vitamins.Every package contains 200ml and provides 260 kcal energy.
  Interventions: Dietary Supplement: enteral nutrition emulsion

INTERVENTIONS:
Dietary Supplement: enteral nutrition emulsion — The patient should drink the oral nutritional supplements according to the estimated energy intake and make a record everyday.The patients will be followed up regularly.
  Arms: nutrition supplementation

SUMMARY:
Insufficient energy intake and systematic inflammation lead to malnutrition in patients with chronic obstructive pulmonary disease (COPD). Nutritional supplementation improves the patients'nutritional status by increasing energy intake and providing anti-inflammatory elements，which can relieve the patients' symptoms and delay the disease progression.

DETAILED DESCRIPTION:
Malnutrition is very common in patients with COPD. The main reasons include short intake of energy and systematic inflammation. In our randomized and controlled clinical trial, patients will be divided into two groups: the experimental group and the control group. Patients in the experimental group will be provided nutritional supplements in addition to usual diet every day for three months and patients in the controlled group with usual diet. According to the changes of patients' body composition, anthropometrics, inflammatory markers, lung function, respiratory muscle function, exercise capacity, degree of dyspnea and health related quality of life(HRQL) after intervention，the nutritional status and inflammation status are assessed, which contributes to the prediction of prognosis. The nutritional supplements is a kind of oral liquid composed of proteins, omega-3 fatty acids, carbohydrate, vitamins, which provides about 260 kcal energy per 200ml. The patients from the interventional group need drink the nutritional supplements according to the estimated energy intake and a record should be made everyday. The patients will be followed up regularly by the researcher.

ELIGIBILITY:
Inclusion Criteria:

Patients from Zhujiang Hospital affiliated from Southern Medical University

Patients aged between 40 and 90 years old

Patients gendered into male or female

Patients with pulmonary function test of FEV1/FVC<70% and FEV1<80% predicted

Patients presenting one or more of the following situations of malnutrition or nutritional risk: BMI <21 kg/m2 (or<23 kg/m2 in patients ≥ 65); unintentional weight loss >10% in the past 6 months; unintentional weight loss >5% in last month; FFMI <15 kg/m2 (women) or <16 kg/m2 (men)

Patients able to answer question

Patient able to eat and drink

Patients who signed informed consent

Exclusion Criteria:

Patients with signs of an airway infection

Patients with malignant disorders

Patients with recent surgery

Patients with gastrointestinal ,cardiovascular diseases,neurological diseases or endocrine disease

Patients with bullae lung

patients treated with oral steroids or immunosuppressors

Patients requiring other nutritional supplements or parenteral nutrition

Patients suffering from acute exacerbation over the previous 4 weeks

Patients with lack of motivation or poor compliance

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-07; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Changes in nutritional status | Before and three months after nutrition supplementation
  Differences in weight,muscle mass(MM),fat mass(FM),free fat mass(FFM),protein，body mass index(BMI),free fat mass index(FFMI) evaluated by bio-impedance measuring technology.
Changes in the serum levels of inflammatory markers | Before and three months after nutrition supplementation
  Changes in the serum levels of tumor necrosis factor-α(TNF-α)、interleukin-6（IL-6）、C-reactive protein(CRP) by laboratory technology.

SECONDARY OUTCOMES:
Changes in pulmonary function | Before and three months after nutrition supplementation
  Differences in forced expiratory volume in first second(FEV1),forced vital capacity(FVC),forced expiratory volume in first second ratio of forced vital capacity(FEV1/FVC) measured by spirometry
Changes in exercise capacity | Before and three months after nutrition supplementation
  Difference in walk distance by six minutes walk test(6MWT)
Changes in anthropometric indexes | Before and three months after nutrition supplementation
  Differences in triceps skinfold thickness（TSF）,mid-arm muscle circumference(MAMC), mid-arm circumference(MAC) measured by tape
Changes in degree of dyspnea | Before and three months after nutrition supplementation
  Difference in dyspnea measured by modified Medical British Research Council（mMRC）
Changes in quality of life score | Before and three months after nutrition supplementation
  Differences in scores measured by Saint George Respiratory Questionaire score
Changes in respiratory muscle function | Before and three months after nutrition supplementation
  Differences in maximal inspiratory pressure（PImax) and maximal expiratory pressure (PEmax) measured by respiratory muscle measurement instrument

CONTACTS AND LOCATIONS:
Overall Officials: Xin Chen, doctor, Principal Investigator — Zhujiang Hospital
Locations (1):
- Zhujiang Hospital,Southern Medical University, Guangzhou, Guangdong, China